CLINICAL TRIAL: NCT01313143
Title: A Prospective, Randomized, Double Blinded, Crossover, Two-treatment, Two-sequence, Short Term Pharmacokinetic, Pharmacodynamic and Tolerability, Single Centre Study to Compare AOP200704 vs. Esmolol in Healthy Subjects.
Brief Title: A Short Term Pharmacokinetic, Pharmacodynamic and Tolerability Study to Compare AOP200704 vs. Esmolol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CPA368-10
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Volunteers; Pharmacokinetics/Dynamics Study
Keywords: AOP200704, Esmolol, Pharmacokinetics, Pharmacodynamics
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOP200704, infusion (Experimental)
  Interventions: Drug: AOP200704
- Esmolol, infusion (Active Comparator)
  Interventions: Drug: Esmolol hydrochloride, infusion

INTERVENTIONS:
Drug: AOP200704 — Comparison of AOP200704 with Esmolol
  Arms: AOP200704, infusion
Drug: Esmolol hydrochloride, infusion — Comparison of AOP200704 with Esmolol
  Arms: Esmolol, infusion

SUMMARY:
Pharmacokinetics, pharmacodynamics and tolerability of AOP200704 infusion is compared to that of Esmolol by measurement of plasma concentrations of AOP200704, esmolol and their metabolites, by assessing the effect of both drugs on dobutamine-induced tachycardia, and by monitoring vital signs, ECG and adverse events.

DETAILED DESCRIPTION:
16 healthy volunteers of both sexes, age 18 to 45 years, will be enrolled. The mean dose necessary to suppress the Dobutamine induced heart rate increase of at least 30 bpm above baseline rate (maximum heart rate app. 110 bpm) by at least 20 bpm will be calculated for AOP200704 and Esmolol and the dose/efficacy relation of both agents to each other will be calculated for the steady state condition. For both drugs the time to reach a decrease of 10 bpm, 20 bpm and the maximum effect will be calculated. In addition the mean time to increase in 10 and 20 bpm and the time to reach maximum heart rate (increase of 30 bpm above baseline or more) after termination of infusion will also be assessed for both drugs. Blood pressure values will be compared for all above mentioned time points where heart rate is assessed for pharmacodynamics.The study will consist of a screening, cross-over 1, cross-over 2 and end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female human subjects, age 18-45 years
* Body weight of at least 50 kg, maximum of 90 kg. Body-mass index 18.5 to 30.0 kg/m2
* Caucasians
* Subjects without clinically relevant abnormalities
* Subjects agreeing to not using any prescription and over the counter medications including vitamins and minerals for 7 days prior to study and during the course of the study
* No drug or alcohol abuse
* Non-smokers, ex smokers and mild smokers

Exclusion Criteria:

* Subjects with history or presence of clinically relevant cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological, psychiatric or skin diseases.
* Subjects with bradycardia (heart rate below 50 bpm), tachycardia (heart rate above 100 bpm), hypotension (systolic blood pressure below 100 mmHg, and/or diastolic blood pressure below 70 mm Hg) at screening, clinically relevant or history of clinically relevant arrhythmias
* Subjects with clinically relevant cardiac supraventricular or ventricular arrhythmias.
* Subjects with atrioventricular block of grade II and III, sick sinus syndrome, sinoatrial block or congestive heart failure
* Participation in a clinical drug study or bioequivalence study 60 days prior to present study.
* History of malignancy or other serious diseases.
* Any contraindication to blood sampling.
* History of i.v. drug abuse.
* Subjects with positive HIV tests, HBsAg or Hepatitis C tests or other acute, subacute or chronic infectious disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics/dynamics | 9 hours

SECONDARY OUTCOMES:
Local tolerability | 9 hours

CONTACTS AND LOCATIONS:
Overall Officials: AOP Study Principal Investigator, Principal Investigator — AOP Contract Clinical Research Facility
Locations (1):
- AOP contract research facility, Pilsen, Czechia